CLINICAL TRIAL: NCT07159035
Title: Flexible Ureteroscopy With a Flexible and Navigable Suction Ureteral Access Sheath Versus Mini-Percutaneous Nephrolithotomy for 1-2 cm Lower Pole Renal Stones: an International, Multicenter, Randomized Non-Inferiority Trial (FLAME Trial)
Brief Title: Flexible Ureteroscopy With a Flexible and Navigable Suction Ureteral Access Sheath Versus Mini-Percutaneous Nephrolithotomy for 1-2 cm Lower Pole Kidney Stones
Acronym: FLAME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Shengjing Hospital (Other); The Third Xiangya Hospital of Central South University (Other); Saint Petersburg State University Hospital (Unknown); Fortune Urology Clinic (Unknown); Zhongda Hospital (Other); Tongji Hospital (Other); The First Affiliated Hospital Hengyang Medical School (Unknown); First Affiliated Hospital of Ningbo University (Network); The Sixth Affiliated Hospital of Guangzhou Medical University (Other); The First Affiliated Hospital of Xiamen University (Other); Dehong People's Hospital (Unknown); People's Hospital of Nanhai District, Foshan (Unknown); Huadu District People's Hospital of Guangzhou (Other); Jiangmen Central Hospital (Other); Baoshan No.2 People's Hospital (Unknown); Guizhou Provincial People's Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Tianjin Medical University Second Hospital (Other); Ankara University (Other)
Responsible Party: Principal Investigator, Guohua Zeng, Vice-president, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ES-2025-181
Record Dates: First submitted 2025-08-28; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Kidney Stones
Keywords: kidney stones; FANS; PCNL; RIRS; flexible ureteroscopy
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio to undergo either FANS-assisted flexible ureteroscopy or mini-percutaneous nephrolithotomy for the treatment of 1-2 cm lower pole renal stones. This is a multicenter, international, randomized, non-inferiority trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding of participants and surgeons is not feasible due to the obvious procedural differences between flexible ureteroscopy with FANS and mini-percutaneous nephrolithotomy. However, radiologists assessing postoperative CT scans will be blinded to treatment allocation. Clinical follow-up assessments will be performed by independent investigators who did not participate in the surgeries. Statistical analysis will also be conducted in a blinded manner, with group assignments concealed from the analyst until data interpretation is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FANS-fURS Group (Experimental): Patients assigned to this group will undergo flexible ureteroscopy with FANS (Flexible endoscopy-Assisted Negative-pressure Suction Sheath). The FANS facilitates direct stone visualization, fragmentation, suction, and removal under controlled pressure conditions.
  Interventions: Procedure: Flexible ureteroscopy with FANS
- mini-PCNL Group (Active Comparator): Patients in this group will receive mini-percutaneous nephrolithotomy (mini-PCNL) via less than 20 Fr percutaneous tracts.
  Interventions: Procedure: Mini-percutaneous nephrolithotomy (mini-PCNL)

INTERVENTIONS:
Procedure: Flexible ureteroscopy with FANS — The FANS with negative-pressure suction, enhancing intrarenal pressure control and fragment evacuation during flexible ureteroscopy.
  Arms: FANS-fURS Group
Procedure: Mini-percutaneous nephrolithotomy (mini-PCNL) — Mini-PCNL is performed under general anesthesia with less than 20 Fr access tract, using rigid nephroscopy and stone fragmentation under direct visualization. Postoperative drainage is provided via nephrostomy or ureteral stent as per protocol.
  Arms: mini-PCNL Group

SUMMARY:
This study, known as the FLAME Trial (Flexible ureteroscopy for Lower pole stones And Mini-pErcutaneous nephrolithotomy), is an international, multicenter, randomized, non-inferiority trial. It aims to compare the effectiveness and safety of flexible ureteroscopy using a flexible and navigable suction ureteral access sheath (FANS) versus mini-percutaneous nephrolithotomy (mini-PCNL) in the treatment of 1-2 cm lower pole kidney stones.

A total of 640 eligible adult patients will be enrolled across 20 high-volume urology centers in China, Russia, Turkey, and India. Participants will be randomly assigned to undergo either FANS-assisted flexible ureteroscopy or mini-PCNL. The primary outcome is the immediate stone-free rate (SFR) assessed by non-contrast CT within 72 hours after surgery. Secondary outcomes include SFR at 1 month, operative time, pain score, length of hospital stay, complication rates, and changes in health-related quality of life.

The goal of this trial is to determine whether the less invasive FANS-assisted approach is non-inferior to mini-PCNL in terms of efficacy, while potentially offering advantages in postoperative recovery and safety.

DETAILED DESCRIPTION:
The FLAME Trial (Flexible ureteroscopy for Lower pole stones And Mini-pErcutaneous nephrolithotomy) is an international, multicenter, prospective, randomized, controlled, non-inferiority study that aims to evaluate the safety and efficacy of flexible ureteroscopy assisted by a Flexible and Navigable Suction Ureteral Access Sheath (FANS) compared with mini-percutaneous nephrolithotomy (mini-PCNL) in the treatment of 1-2 cm lower pole renal stones.

This trial will enroll 640 patients from 20 urology centers with substantial experience in endoscopic stone surgery, including hospitals in China, Russia, Turkey, and India. Eligible participants will be randomly assigned in a 1:1 ratio to either the FANS-assisted flexible ureteroscopy group or the mini-PCNL group. All patients will undergo preoperative imaging, intraoperative standardization, and postoperative follow-up according to the study protocol.

The primary endpoint is the stone-free rate (SFR) within 72 hours postoperatively, evaluated by non-contrast-enhanced computed tomography (NCCT). Secondary endpoints include SFR at 1 month, operative time, length of hospital stay, postoperative pain (measured by VAS score), complication rates (graded by Clavien-Dindo classification), changes in renal function, and health-related quality of life (HRQoL).

The FANS, developed to improve irrigation control and active stone fragment suction during flexible ureteroscopy, may provide better visualization, reduce intrarenal pressure, and shorten operative time. By directly comparing FANS-assisted fURS with mini-PCNL, the trial seeks to determine whether a less invasive method can achieve comparable outcomes in terms of stone clearance and complication rates.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18-75 years;
2. American Society of Anesthesiology (ASA) score 1-3;
3. Lower pole renal stones-single or multiple-with a maximal diameter of 1-2 cm confirmed by CT;
4. Ability to provide written informed consent and adhere to trial requirements.

Exclusion Criteria:

1. Significant urinary tract anatomical anomalies (e.g. horseshoe kidney, ileal conduit);
2. Stones located within a calyceal diverticulum;
3. History of open nephrolithotomy or ureterolithomy (due to resultant intrarenal anatomical distortion);
4. Absolute contraindications to either FANS-f-URS or mini-PCNL, including:

   * Uncorrectable coagulopathy;
   * Active, uncontrolled urinary tract infection;
   * Severe cardiopulmonary disease precluding safe general anesthesia (e.g. decompensated heart failure, refractory COPD);
   * Pregnancy;
   * Inability to tolerate lithotomy or prone positioning;
5. Inability to understand or complete trial documentation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Immediate Stone-Free Rate (SFR) | 72 hours after surgery
  Stone-free status will be evaluated using non-contrast-enhanced computed tomography (NCCT) performed within 72 hours after surgery. Stone-free is defined as the absence of residual stone fragments or presence of clinically insignificant fragments ≤2 mm.

SECONDARY OUTCOMES:
Final Stone-Free Rate (SFR) at 1 Month | 1 month after surgery
  Assessed by low-dose CT scan. Patients with no residual stones or with residual fragments ≤2 mm are defined as stone-free.
Operative Time | Intraoperative
  For the FANS-fURS group, operative time is defined as the duration from insertion of the endoscope into the urethra to completion of stent placement.
  For the mini-PCNL group, it is defined as the time from retrograde placement of the ureteric catheter to nephrostomy tube placement or percutaneous access removal.
Postoperative Pain Level | Within 24 hours after surgery.
  Evaluated using the 10-point Visual Analog Scale (VAS), where 0 indicates no pain and 10 indicates worst pain.
Length of Hospital Stay | From the day of surgery until the day of discharge, assessed up to 30 days postoperatively.
  From surgery to discharge.
Complication Rate Within 1 Month | 1 month after surgery.
  All postoperative complications will be recorded and graded using the Clavien-Dindo classification system.
Change in Quality of Life Score | Baseline and 1 month after surgery.
  Assessed using the Wisconsin Stone Quality of Life (WISQOL) questionnaire before surgery and at 1-month follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to institutional policy restrictions and data privacy considerations.

REFERENCES:
- [Background] Skolarikos A, Geraghty R, Somani B, Tailly T, Jung H, Neisius A, Petrik A, Kamphuis GM, Davis N, Bezuidenhout C, Lardas M, Gambaro G, Sayer JA, Lombardo R, Tzelves L. European Association of Urology Guidelines on the Diagnosis and Treatment of Urolithiasis. Eur Urol. 2025 Jul;88(1):64-75. doi: 10.1016/j.eururo.2025.03.011. Epub 2025 Apr 22. PMID 40268592
- [Derived] Zhu W, Zhong J, Wang K, Yin G, Leung CH, Gadzhiev N, Gokce MI, Kalathia J, Gauhar V, Zhang G, Wu G, Li M, Fang L, Zeng S, Bai P, Li J, Zhao Z, Xi M, Mai X, Duan X, Jiang K, Cao J, Meng X, Liu S, Aloyan A, Yuan P, Zhu X, Huang T, Xing J, Du J, Wu W, Ma J, Zhong W, Zhao Z, Liu Y, Ng CF, de la Rosette J, Somani B, Qi S, Zeng G, Yuen SKK. Flexible ureteroscopy with a flexible and navigable suction ureteral access sheath versus mini-percutaneous nephrolithotomy for 1-2 cm lower pole renal stones: Protocol for an international, multicentre, randomized non-inferiority trial (FLAME trial). BJUI Compass. 2025 Nov 29;6(12):e70114. doi: 10.1002/bco2.70114. eCollection 2025 Dec. PMID 41323963